CLINICAL TRIAL: NCT04454905
Title: A Single-arm Phase II Study to Evaluate Camrelizumab in Combination With Apatinib in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Camrelizumab in Combination With Apatinib in Advanced ICC: A Single-arm Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-098-01
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — camrelizumab; Injections; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combination with Apatinib (Experimental): Camrelizumab 200mg, every 3 weeks, intravenous infused. Apatinib 250mg, once a day, orally. Until progression or unacceptable toxicity events develop.
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab (Jiangsu HengRui Medicine Co., Ltd.) is a recombinant anti-human PD-1 IgG4 monoclonal antibody.
  Other Names: Camrelizumab for Injection
Drug: Apatinib — Apatinib is a novel angiogenesis inhibitor vascular endothelial growth factor 2.
  Other Names: Rivoceranib

SUMMARY:
This is a single arm, open-label, non-randomized and single-center phase II clinical study, to evaluate the safety, tolerance, and efficacy of Camrelizumab in combination with Apatinib in patients with advanced intrahepatic cholangiocarcinoma (ICC).

DETAILED DESCRIPTION:
It is estimated that 50 patients who met the study criteria will be enrolled in 3 years and treated with Camrelizumab plus Apatinib in SYSUCC. The investigators will follow up and collect subjects' data to evaluate the efficacy and safety of treatment, including objective response rate (ORR) and Progression-free Survival (PFS) and Overall Survival (OS), until disease progression or death. Histopathology and multi-omics data analysis will be used to explore potential biomarkers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed advanced ICC, or combined hepatocellular and cholangiocarcinoma (cHCC-CC, composition of cholangiocarcinoma >50%). nonresectable or metastatic cholangiocarcinoma and are not eligible for curative resection, transplantation, or ablative therapies.
* Have at least one measurable lesion (in accordance with RECIST v1.1); the measurable lesion has a long diameter ≥ 10 mm or lymphadenopathy has a short diameter ≥ 15 mm in spiral CT scan.
* Child-Pugh Class: Grade A
* ECOG-PS score 0 or 1
* Life Expectancy of at least 3 months
* Have the required screening laboratory values

Exclusion Criteria:

* Extrahepatic cholangiocarcinoma (EHCC) and primary liver cancer. other active malignant tumors except for ICC within 3 years or simultaneously. Cured localized tumor, for example, basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situs of cervix, breast cancer in situ may be enrolled.
* Any active autoimmune disease or history of autoimmune disease and expected recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects that can be controlled with hormone replacement therapy only can be enrolled]); subjects with skin diseases that does no need systemic treatment, for example, leukoderma, psoriasis, alopecia, those with controlled type I diabetes by insulin or those with asthma that has been completely resolved in childhood and with no need of any intervention can be enrolled; while subjects with asthma who need bronchodilator for medical intervention cannot be enrolled;
* Use of strong CYP3A4/CYP2C19 inducers, including rifampicin (and its analogues) and St. John's Wort, or strong CYP3A4/CYP2C19 inhibitors within two weeks prior to signing informed consent form.
* Previous treatment with other immune checkpoint inhibitors (include PD-1 antibody or other immunotherapy against PD-1/PD-L1), or previous use of Apatinib.
* Known history of serious allergy to any monoclonal antibody or Apatinib.
* Inability or unwilling to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption.
* Previous or current presence of metastasis to central nervous system.
* Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; oral or intravenous therapeutic antibiotics within two weeks prior to the start of study treatment (for example, subjects who are given with preventive antibiotics for prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for participation in the study);
* Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring concomitant therapy, with serious laboratory examination abnormality, with family or social factors, that may affect subject's safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Three years
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Three years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Overall Survival (OS) | Three years
  Duration from the date of initial treatment to the date of death due to any cause.
Disease Control Rate (DCR) | Two years
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Duration of Response (DoR) | Two years
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Time to Progression (TTP) | Two years
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1)
Adverse events (AE) | Two years
  Any adverse events related with treatment drugs and details include adverse events type, frequency and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Minshan Chen, MD., PhD., Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Li Xu, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong